CLINICAL TRIAL: NCT05059938
Title: Promoting the Use of Free Smartphone App (MyFitnessPal) for Weight Loss by Primary Care Provider in Overweight Patients: A Randomized Controlled Pilot Study
Brief Title: MyFitnessPal Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator changed positions
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Kristin Simmons Bennie, Physician Primary Care, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0907
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Weight Reduction
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyFitnessPal user (Experimental): Patients will be shown how to download and use MyFitnessPal onto the patient's smartphone. The patient will be asked to use the application to aid in the patient's weight loss plan over up to six months.
  Interventions: Behavioral: MyFitnessPal user
- Traditional Weight Loss Counseling (No Intervention): Patients will be given traditional weight loss counseling from the physician and monitored over up to six months.

INTERVENTIONS:
Behavioral: MyFitnessPal user — Patients will be counseled on how to use the MyFitnessPal application to help with the patient's weight loss goals. The physician will monitor the patient's weight, blood pressure, and waist circumference over up to a six month period with visits at 1, 3, and 6 months. Patients will be asked about the patient's use of the application at the end of the study.
  Arms: MyFitnessPal user

SUMMARY:
This project is studying whether patients who use MyFitnessPal as an aid to weight loss have more success than patients who are only given traditional medical guidance from the patient's physician.

DETAILED DESCRIPTION:
Patients will be given a survey determining the patient's eligibility to be part of the study. Based on the results patients will be consented and then randomized into two arms. The intervention group will download MyFitnessPal onto the patient's smartphone and given guidance on how to use the application in order to help with weight loss. The control group will receive traditional weight loss counseling from the physician. Both groups will have measurement recorded for weight, blood pressure, and waist circumference at the patient's initial visit. All patients will be asked to return to the clinic at no cost to the patient to have measurements recorded for the patient's weight, blood pressure, and waist circumference at 1 month, 3 months, and 6 months after the patient's initial visit. At the conclusion of the study, patients who were in the intervention group will be asked to take a final survey regarding the patient's use of the MyFitnessPal application.

ELIGIBILITY:
Inclusion Criteria:

* BMI>/= 25
* Have a smart phone
* Patient is willing to lose weight

Exclusion Criteria:

* Do not have a smart phone
* pregnant (current, planned, or previous pregnancy within 6 months)
* have already seen a nutritionist
* on weight loss medication
* using outside weight loss programs
* lack interest in weight loss
* hemodialysis patient
* has a life expectancy less than 6 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Weight Loss | 1-6 months
  Weight will be measured in pounds and recorded at each visit

SECONDARY OUTCOMES:
Change in Waist Circumference | 1-6 months
  Waist Circumference will be measured in centimeters and recorded at each visit
Change in Blood Pressure | 1-6 months
  Blood pressure will be measured and recorded at each visit

OTHER OUTCOMES:
Pre-Screen survey | First visit
  Patients will be asked about willingness to participate in weight loss and other inclusion/exclusion questions
Post intervention survey | 3 to 6 months
  Patients will be asked about overall use of the application and how it affected weight loss.

IPD SHARING:
Plan to Share IPD: No